CLINICAL TRIAL: NCT02635516
Title: Treatment of Mild and Moderate Traumatic Brain Injury in Veterans Using Near-Infrared Phototherapy
Brief Title: Traumatic Brain Injury in Veterans and Near-Infrared Phototherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cerehealth Corp. (Industry)
Collaborators: Tug McGraw Foundation (Unknown); Colorado Neurological Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014.01.01
Record Dates: First submitted 2015-12-15; First posted 2015-12-21 (Estimated); Last update posted 2015-12-21 (Estimated); Status verified 2015-12

CONDITIONS: TBI (Traumatic Brain Injury)
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental): Only one arm was used and this arm received Near-Infrared Phototherapy.
  Interventions: Device: Near-Infrared Phototherapy

INTERVENTIONS:
Device: Near-Infrared Phototherapy — The In Light Wellness Systems Near-Infrared Phototherapy Device (manufactured by In Light Wellness Systems, Inc.) contains alternating rows of 402 red (640 nm) and infrared (880 nm) light-emitting diodes embedded in 2 neoprene pads. One pad circles the skull, providing 720 Joules/min, and the other pad covers the top of the head, providing 360 joules/min. For each treatment session, the "A" setting on the 3-port controller is utilized, which runs approximately 6.7 min of 73 Hz, 587 Hz, and 1175 Hz in an automated sequential manner. No other interventions were utilized.
  Other Names: Polychromatic Light Therapy

SUMMARY:
This is a proof-of-concept study designed to demonstrate whether increases in cerebral blood flow, improvements in brain functioning, and reductions in symptomology associated with traumatic brain injury (TBI) can result from treatments consisting of near-infrared phototherapy (NIR).

DETAILED DESCRIPTION:
The incidence of traumatic brain injury is widespread. The Centers for Disease Control estimate that 1.7 million TBIs occur each year and that TBI is a contributing factor in about 30% of all injury-related deaths. In addition, about 75% of these TBIs are concussions, or mild TBIs (mTBI). However, such concussions, especially multiple concussions that occur over time, are not harmless. The damage of even mild TBI can potentially lead to neuropsychiatric sequelae. Moreover, injury to the brain can worsen over time depending on the degree of inflammatory response and the areas of injury. TBI induces a number of neuropathological changes like aggregation of beta amyloid and tau proteins along with neuroinflammatory changes that resemble the pathology of degenerative diseases.

For many of our returning Veterans, improvised explosive devices (IEDs) have been the cause of these TBIs. For example, data from the Defense Manpower Data Center indicates that as of October 3, 2011, explosive devices have been responsible for an estimated two-thirds or more of the battlefield injuries in Iraq; of the 46,532 warriors wounded in Operations Enduring Freedom and Iraqi Freedom, 30,347 were wounded by explosive devices, many of which were IEDs. Most of these injuries involved concussive brain injury. While current estimates are that 15-19% of all returning Warfighters have a history of acute concussion or TBI during their tour(s) of duty. It has been noted that "22.8% of a Brigade Combat Team returned from Iraq with confirmed deployment-acquired traumatic brain injury."

Currently, there are no effective treatments for reversing or reducing the brain damage following TBI. Confounding the situation further, the symptoms of TBI can often overlap with those of post-traumatic stress disorder (PTSD) such as headache, dizziness, irritability, memory impairment, delayed problem solving, slowed reaction time, fatigue, visual disturbances, sleep disturbances, sensitivity to light and noise, impulsivity, judgment problems, emotional outbursts, depression, and anxiety. In addition, the rates of depression, anxiety, and other psychological symptoms are markedly elevated in TBI survivors, based on studies involving large samples of patients. As a result of this complexity and overlap of symptoms between TBI, PTSD, and depression, a clear diagnosis of TBI can be challenging, which can lead to misdirected treatment efforts and hamper the ability to accurately assess treatment response.

Multiple published research studies have validated the healing mechanisms of NIR, which can be delivered via light-emitting diodes (LED). NIR phototherapy has been used extensively for wound healing of soft tissue, for increasing circulation, for the treatment of pain and for specific conditions such as hair growth and carpal tunnel syndrome.

The mechanism of action that is central to the healing effect of NIR is increased blood circulation via the release of nitric oxide from red blood cells. Local increases in nitric oxide increase blood flow through arteries, veins and lymphatic ducts. Increased return of flow from treated sites helps to diminish intracellular acidosis that could alter mitochondrial membrane potential(s). This hypothesis holds that when blood flow is adequate, it provides a sufficient amount of oxygen and glucose to cells for adenosine triphosphate (ATP) generation by mitochondria. However, even a modest decrease in regional or global blood flow in the brain, such as that seen in TBI, will limit the amount of glucose and oxygen delivered to neurons. Restoring blood flow levels in damaged regions of the brain thus restores the necessary levels of glucose and oxygen required for ATP generation and proper neuronal functioning.

In addition, nitric oxide stimulates angiogenesis and increased numbers of capillaries will aid in increasing blood flow (and oxygen and glucose) in injured areas of the brain where blood flow was subnormal. This effect contributes to enhanced mitochondrial function. The 1998 Nobel Prize for physiology was awarded to Furchgott, Ignarroand, and Murad for their discovery that nitric oxide acts as a signaling molecule and activates an enzyme, guanylate cyclase (GC), which is necessary for subsequent vasodilation.

Finally, nitric oxide is an effective analgesic; it appears to reduce pain either by reversing local ischemia or directly in a manner akin to the analgesic effect of morphine. In the latter case, nitric oxide helps to regulate membrane potential via alterations in the activity of the ATP dependent potassium channel. This effect may be mediated by activated GC and subsequent phosphorylation of the potassium channel.

Due to its capacity to non-invasively penetrate the skull, NIR has been safely used since the late 1970s for the determination of cerebral blood flow and oxygen levels in brain injured adults, post-stroke patients, and in pediatric patients. Furthermore, transcranial NIR has been shown to increase cortical perfusion and is associated with clinical improvement in human subjects with traumatic brain injury, neurodegenerative disease, and depression. The NIR device for this study is FDA cleared (510K; K101894) for increasing circulation and reducing pain.

ELIGIBILITY:
Inclusion Criteria:

1. Participant is a military veteran.
2. Able to read and sign the Informed Consent.
3. Clinical history and diagnosis of TBI.
4. Incident of TBI occurred at least 18 months or more prior to enrollment.
5. Participant is willing and able to follow protocols for SPECT imaging procedure.
6. SPECT scan shows evidence of TBI.

Exclusion Criteria:

1. Participant is not a military veteran.
2. Unable to read or sign the Informed Consent.
3. No prior clinical indications of TBI.
4. Participant is unwilling or unable to follow protocols for SPECT imaging procedure.
5. SPECT scan shows no evidence of TBI.
6. SPECT scan shows evidence of TBI but with significant comorbid neurological condition(s), which include active suicidal or homicidal ideation, psychosis, or repetitive expression of delusional ideation. In addition, any other psychiatric, neurological, orthopedic or cardiopulmonary condition that would preclude the ability of the subject to lie still for scan acquisition for 25-30 minutes and/or participate fully in the treatment regimen will result in exclusion from the study.

Ages: 21 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2014-04; Primary Completion 2015-03 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Change in Cerebral Blood Flow | Time1: Resting SPECT brain scan 2-14 days pre-treatment; Time2: Resting SPECT brain scan 1-4 weeks post-treatment.
  Single photon emission computed tomography (SPECT). To obtain this outcome measure, at pre- and post-treatment, a resting SPECT brain scan is performed as follows. Patient is placed in a comfortable reclining chair in a quiet room and an IV is started. Patient is allowed to acclimate in a quiet, semi-darkened room with eyes open and sound-dampening headphones on for 15 min, in accordance with the 2014 American College of Radiology Practice Guidelines. After 15 min., a dose of approximately 30 millicuries of Technetium-99m radiotracer is injected. SPECT scan is performed 60 min following injection by using a Siemens Symbia E SPECT gamma camera with low-energy high-resolution parallel hole collimators.
Change in TBI Symptoms | T1: 2-14 days prior to pre-treatment concentration brain scan; T2: 1-4 weeks post-treatment.
  Self-report TBI symptoms inventory composed of Likert-type items constructed to measure both frequency and intensity of 15 TBI symptoms.
Change in Cognitive Functioning | T1: 2-14 days prior to pre-treatment concentration brain scan; T2: 1-4 weeks post-treatment.
  Neuropsychological testing focused on the cognitive abilities frequently affected by TBI. Includes subscales of the Wechsler Adult Intelligence Scale IV.

SECONDARY OUTCOMES:
Change in Cognitive Functioning 2 | T1: 2-14 days prior to pre-treatment SPECT brain scan; T2: 1-4 weeks post-treatment.
  Neuropsychological testing focused on the cognitive abilities frequently affected by TBI. Includes subscales of the California Verbal Learning Test II.
Change in Cognitive Functioning 3 | T1: 2-14 days prior to pre-treatment SPECT brain scan; T2: 1-4 weeks post-treatment.
  Neuropsychological testing focused on the cognitive abilities frequently affected by TBI. Includes the Trail Making Test B.

CONTACTS AND LOCATIONS:
Overall Officials: Fred Grover, Jr., M.D., Principal Investigator — RevolutionaryMD

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant relevant demographic data will be reported. De-identified individual data analyses will be reported.

REFERENCES:
- [Background] Abdel-Dayem HM, Abu-Judeh H, Kumar M, Atay S, Naddaf S, El-Zeftawy H, Luo JQ. SPECT brain perfusion abnormalities in mild or moderate traumatic brain injury. Clin Nucl Med. 1998 May;23(5):309-17. doi: 10.1097/00003072-199805000-00009. PMID 9596157
- [Background] Fann JR, Burington B, Leonetti A, Jaffe K, Katon WJ, Thompson RS. Psychiatric illness following traumatic brain injury in an adult health maintenance organization population. Arch Gen Psychiatry. 2004 Jan;61(1):53-61. doi: 10.1001/archpsyc.61.1.53. PMID 14706944
- [Background] Hoge CW, Castro CA, Messer SC, McGurk D, Cotting DI, Koffman RL. Combat duty in Iraq and Afghanistan, mental health problems and barriers to care. US Army Med Dep J. 2008 Jul-Sep:7-17. PMID 20088060
- [Background] Jacobs A, Put E, Ingels M, Put T, Bossuyt A. One-year follow-up of technetium-99m-HMPAO SPECT in mild head injury. J Nucl Med. 1996 Oct;37(10):1605-9. PMID 8862291
- [Background] Jorge RE, Robinson RG, Moser D, Tateno A, Crespo-Facorro B, Arndt S. Major depression following traumatic brain injury. Arch Gen Psychiatry. 2004 Jan;61(1):42-50. doi: 10.1001/archpsyc.61.1.42. PMID 14706943
- [Background] Kashluba S, Hanks RA, Casey JE, Millis SR. Neuropsychologic and functional outcome after complicated mild traumatic brain injury. Arch Phys Med Rehabil. 2008 May;89(5):904-11. doi: 10.1016/j.apmr.2007.12.029. PMID 18452740
- [Background] Kennedy JE, Jaffee MS, Leskin GA, Stokes JW, Leal FO, Fitzpatrick PJ. Posttraumatic stress disorder and posttraumatic stress disorder-like symptoms and mild traumatic brain injury. J Rehabil Res Dev. 2007;44(7):895-920. doi: 10.1682/jrrd.2006.12.0166. PMID 18075948
- [Background] Langlois JA, Rutland-Brown W, Wald MM. The epidemiology and impact of traumatic brain injury: a brief overview. J Head Trauma Rehabil. 2006 Sep-Oct;21(5):375-8. doi: 10.1097/00001199-200609000-00001. PMID 16983222
- [Background] Lew HL. Rehabilitation needs of an increasing population of patients: Traumatic brain injury, polytrauma, and blast-related injuries. J Rehabil Res Dev. 2005 Jul-Aug;42(4):xiii-xvi. No abstract available. PMID 16320135
- [Background] Nawashiro H, Wada K, Nakai K, Sato S. Focal increase in cerebral blood flow after treatment with near-infrared light to the forehead in a patient in a persistent vegetative state. Photomed Laser Surg. 2012 Apr;30(4):231-3. doi: 10.1089/pho.2011.3044. Epub 2011 Nov 2. PMID 22047598
- [Background] Schiffer F, Johnston AL, Ravichandran C, Polcari A, Teicher MH, Webb RH, Hamblin MR. Psychological benefits 2 and 4 weeks after a single treatment with near infrared light to the forehead: a pilot study of 10 patients with major depression and anxiety. Behav Brain Funct. 2009 Dec 8;5:46. doi: 10.1186/1744-9081-5-46. PMID 19995444
- [Background] Vaishnavi S, Rao V, Fann JR. Neuropsychiatric problems after traumatic brain injury: unraveling the silent epidemic. Psychosomatics. 2009 May-Jun;50(3):198-205. doi: 10.1176/appi.psy.50.3.198. PMID 19567758